CLINICAL TRIAL: NCT04394780
Title: Pilot Study to Determine Whether Cooled Peritoneal Dialysis Fluid Confers Cardio-Protective Effects
Brief Title: Peritoneal Dialysis Fluid Cooling and Cardio-Protective Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 107280
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Dialysis; Complications
Keywords: cooling; peritoneal dialysis; myocardial perfusion; myocardial heterogeneity
MeSH Terms: interventions — Cool-Down Exercise

STUDY DESIGN:
Intervention Model Description: Every patient underwent peritoneal dialysis at 37 C and then at 32 C one week after.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peritoneal dialysis at 37 C (No Intervention): Patients underwent peritoneal dialysis with the standard temperature.
- Peritoneal dialysis at 32 C (Active Comparator): Patients started on continuous ambulatory peritoneal dialysis using a peritoneal dialysate cooled to between 32-33 degrees centigrade, at a pre-determined and precisely controlled temperature for the 4 hour duration treatment.
  Interventions: Procedure: cooling

INTERVENTIONS:
Procedure: cooling — First, patients underwent peritoneal dialysis (PD) at 37 C (standard temperature) and then patients underwent PD cooling. After each PD session, the patient had a CT scan for the study team to study myocardial perfusion at rest and after introduction of a pharmacological stressor.
  Arms: Peritoneal dialysis at 32 C

SUMMARY:
The study team aimed to investigate the relationship between occlusive coronary artery disease, myocardial perfusion, and peritoneal dialysate temperature. In addition, the study team aimed to identify how abnormal myocardial perfusion in peritoneal dialysis (PD) patients is related to occlusive coronary artery disease, to identify factors associated with occlusive coronary artery disease in end-stage renal failure patients on PD. Finally, the study team identified factors associated with PD induced cardiac injury in end-stage renal failure patients on this dialysis modality.

In order to assess the patients response to physiological stress and the functional relevance of their coronary artery disease, patients underwent assessment using dual energy contrast enhanced (DCE) CT assessment of coronary arteries and myocardial perfusion. An initial CT scan with administration of contrast established baseline information regarding the extent of coronary artery disease, fibrosis, and myocardial perfusion at rest. Following this, patients underwent pharmacological stress with the administration of adenosine and a repeat CT scan established the response to stress in terms of myocardial perfusion. On the second study visit patients were started on C-CAPD using peritoneal dialysate cooled to between 32-33 degrees centigrade, at a pre-determined and precisely controlled temperature for the 4 hour duration of C-CAPD. Subsequently, patients were injected with a pharmacological stressor in the form of adenosine. They then underwent DCE CT assessment of coronary arteries and myocardial perfusion as done in the first visit. The second CT scan took place following a PD dwell.

ELIGIBILITY:
Inclusion Criteria:

* Patients having peritoneal dialysis treatment at least 6 times per week at home and followed at the London Health Sciences Centre
* Male and female, age=16 years old
* Patients listed for renal transplantation
* Residual renal function less than or equal to 750 mls per 24 hour period

Exclusion Criteria:

* Not meeting inclusion criteria
* Previous adverse reaction to intravenous contrast
* Allergy to adenosine - Patients with significant residual renal function (greater than 750mL/24 hours)
* Exposure to peritoneal dialysis for <90 days prior to recruitment
* Ongoing spontaneous bacterial peritonitis (SBP)
* Severe heart failure (New York Heart Association grade IV) - Cardiac transplant recipients
* Mental incapacity to consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Correlation between occlusive coronary artery disease and myocardial perfusion | The day of study visit 1, lasting for approximately 2 hours
  Investigate the correlation between occlusive coronary artery disease, myocardial perfusion, and peritoneal dialysate temperature. Patients will have a CT scan to measure perfusion (mL/min/g) after peritoneal dialysis
Correlation between occlusive coronary artery disease and myocardial perfusion | The day of study visit 2, lasting for approximately 6 hours
  Investigate the correlation between occlusive coronary artery disease, myocardial perfusion and peritoneal dialysate temperature. Patients will have a CT scan to measure perfusion (mL/min/g) after peritoneal dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No
We don't share participant data with other researchers except our team

REFERENCES:
- [Result] Kalantar-Zadeh K, Block G, Humphreys MH, Kopple JD. Reverse epidemiology of cardiovascular risk factors in maintenance dialysis patients. Kidney Int. 2003 Mar;63(3):793-808. doi: 10.1046/j.1523-1755.2003.00803.x. PMID 12631061
- [Result] Burton JO, Jefferies HJ, Selby NM, McIntyre CW. Hemodialysis-induced cardiac injury: determinants and associated outcomes. Clin J Am Soc Nephrol. 2009 May;4(5):914-20. doi: 10.2215/CJN.03900808. Epub 2009 Apr 8. PMID 19357245
- [Result] Boon D, Bos WJ, van Montfrans GA, Krediet RT. Acute effects of peritoneal dialysis on hemodynamics. Perit Dial Int. 2001 Mar-Apr;21(2):166-71. PMID 11330561
- [Result] Drueke TB, Massy ZA. Atherosclerosis in CKD: differences from the general population. Nat Rev Nephrol. 2010 Dec;6(12):723-35. doi: 10.1038/nrneph.2010.143. Epub 2010 Oct 26. PMID 20978469
- [Result] McIntyre CW. Effects of hemodialysis on cardiac function. Kidney Int. 2009 Aug;76(4):371-5. doi: 10.1038/ki.2009.207. Epub 2009 Jun 10. PMID 19516249
- [Result] Ragosta M, Samady H, Isaacs RB, Gimple LW, Sarembock IJ, Powers ER. Coronary flow reserve abnormalities in patients with diabetes mellitus who have end-stage renal disease and normal epicardial coronary arteries. Am Heart J. 2004 Jun;147(6):1017-23. doi: 10.1016/j.ahj.2003.07.029. PMID 15199350
- [Result] Selby NM, Fialova J, Burton JO, McIntyre CW. The haemodynamic and metabolic effects of hypertonic-glucose and amino-acid-based peritoneal dialysis fluids. Nephrol Dial Transplant. 2007 Mar;22(3):870-9. doi: 10.1093/ndt/gfl654. Epub 2006 Nov 22. PMID 17121785
- [Result] Verbeke F, Van Biesen W, Pletinck A, Van Bortel LM, Vanholder R. Acute central hemodynamic effects of a volume exchange in peritoneal dialysis. Perit Dial Int. 2008 Mar-Apr;28(2):142-8. PMID 18332449
- [Result] Selby NM, Fonseca S, Hulme L, Fluck RJ, Taal MW, McIntyre CW. Automated peritoneal dialysis has significant effects on systemic hemodynamics. Perit Dial Int. 2006 May-Jun;26(3):328-35. PMID 16722025
- [Result] Barnes E, Dutka DP, Khan M, Camici PG, Hall RJ. Effect of repeated episodes of reversible myocardial ischemia on myocardial blood flow and function in humans. Am J Physiol Heart Circ Physiol. 2002 May;282(5):H1603-8. doi: 10.1152/ajpheart.00786.2001. PMID 11959621
- [Result] McIntyre CW, Burton JO, Selby NM, Leccisotti L, Korsheed S, Baker CS, Camici PG. Hemodialysis-induced cardiac dysfunction is associated with an acute reduction in global and segmental myocardial blood flow. Clin J Am Soc Nephrol. 2008 Jan;3(1):19-26. doi: 10.2215/CJN.03170707. Epub 2007 Nov 14. PMID 18003765
- [Result] Burton JO, Jefferies HJ, Selby NM, McIntyre CW. Hemodialysis-induced repetitive myocardial injury results in global and segmental reduction in systolic cardiac function. Clin J Am Soc Nephrol. 2009 Dec;4(12):1925-31. doi: 10.2215/CJN.04470709. Epub 2009 Oct 1. PMID 19808220
- [Result] Erlinge D. A Review of Mild Hypothermia as an Adjunctive Treatment for ST-Elevation Myocardial Infarction. Ther Hypothermia Temp Manag. 2011;1(3):129-41. doi: 10.1089/ther.2011.0008. PMID 24717042
- [Result] Gotberg M, Olivecrona GK, Engblom H, Ugander M, van der Pals J, Heiberg E, Arheden H, Erlinge D. Rapid short-duration hypothermia with cold saline and endovascular cooling before reperfusion reduces microvascular obstruction and myocardial infarct size. BMC Cardiovasc Disord. 2008 Apr 10;8:7. doi: 10.1186/1471-2261-8-7. PMID 18402663
- [Result] Chopp M, Knight R, Tidwell CD, Helpern JA, Brown E, Welch KM. The metabolic effects of mild hypothermia on global cerebral ischemia and recirculation in the cat: comparison to normothermia and hyperthermia. J Cereb Blood Flow Metab. 1989 Apr;9(2):141-8. doi: 10.1038/jcbfm.1989.21. PMID 2921288
- [Result] Jefferies HJ, Burton JO, McIntyre CW. Individualised dialysate temperature improves intradialytic haemodynamics and abrogates haemodialysis-induced myocardial stunning, without compromising tolerability. Blood Purif. 2011;32(1):63-8. doi: 10.1159/000324199. Epub 2011 Feb 24. PMID 21346338
- [Result] Odudu A, Eldehni MT, McCann GP, McIntyre CW. Randomized Controlled Trial of Individualized Dialysate Cooling for Cardiac Protection in Hemodialysis Patients. Clin J Am Soc Nephrol. 2015 Aug 7;10(8):1408-17. doi: 10.2215/CJN.00200115. Epub 2015 May 11. PMID 25964310
- [Result] Eldehni MT, Odudu A, McIntyre CW. Randomized clinical trial of dialysate cooling and effects on brain white matter. J Am Soc Nephrol. 2015 Apr;26(4):957-65. doi: 10.1681/ASN.2013101086. Epub 2014 Sep 18. PMID 25234925